CLINICAL TRIAL: NCT04067791
Title: A Randomized, Double-blind, Comparator-controlled, Cross-over Study to Investigate the Pharmacokinetics of Prolonged-release Melatonin Compared to Standard, Immediate-release Melatonin in Healthy Adults
Brief Title: A Study to Investigate the Pharmacokinetics of Prolonged-release Melatonin Compared to Standard, Immediate-release Melatonin in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmavite LLC (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 19MPHP
Record Dates: First submitted 2019-08-19; First posted 2019-08-26 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Healthy
Keywords: Healthy; Adult; Melatonin; Pharmacokinetic; Absorption; prolonged-release; immediate-release

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prolonged-Release melatonin then Immediate-release melatonin (Experimental)
  Interventions: Dietary Supplement: Prolonged-Release Melatonin; Dietary Supplement: Immediate-Release Melatonin
- Immediate-Release Melatonin then Prolonged-Release Melatonin (Experimental)
  Interventions: Dietary Supplement: Prolonged-Release Melatonin; Dietary Supplement: Immediate-Release Melatonin

INTERVENTIONS:
Dietary Supplement: Prolonged-Release Melatonin — 4.47 mg melatonin in a bi-layer prolonged-release capsule
Dietary Supplement: Immediate-Release Melatonin — 4.47 mg melatonin in a standard release bi-layer capsule

SUMMARY:
A study comparing the pharmacokinetics of prolonged-release melatonin versus standard, immediate-release melatonin. Multiple blood draws over a 10-hour period will be analysed to determine the area under the curve, time to peak concentration, peak concentration, absorption rate constant, elimination rate constant, absorption half-life, and elimination half-life. Vital signs, hematology parameters, clinical chemistry parameters, and incidence of adverse events are also analysed.

ELIGIBILITY:
Inclusion Criteria:

1. Females and males between 18 and 65 years of age at screening
2. BMI between 18.5 to 29.9 kg/m2, inclusive
3. Female participant is not of child-bearing potential, defined as females who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, total endometrial ablation) or have been post-menopausal (natural or surgically) for at least 1 year prior to screening Or, Females of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. Acceptable methods of birth control include: e. Non-hormonal intrauterine devices f. Double-barrier method g. Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s) h. Vasectomy of partner at least 6 months prior to screening
4. Male participants must agree to the use of condoms unless partner is using an acceptable form of female contraception as defined in Inclusion #3 or a form of hormonal birth control during the study treatment period and for at least 7 days after completion of the study
5. Have a regular sleep-wake cycle with a bedtime between 9:00 pm and 12:00 am and receive between 7 and 8 hours of sleep for at least 3 weeks
6. Agrees to maintain current sleep schedule throughout study
7. Agrees to maintain current level of physical activity and diet throughout the study
8. Agrees to comply with all study procedures
9. Agrees to consume standardized meals during Visits 2 and 3
10. Agrees to avoid caffeine intake 24 hours prior to Visits 2 and 3
11. Agrees to avoid alcohol intake 24 hours prior to Visits 2 and 3
12. Healthy as determined by medical history, laboratory results, and physical exam as assessed by QI
13. Agrees to provide informed written consent

Exclusion Criteria:

1. Women who are pregnant, breastfeeding or planning to become pregnant during the course of the trial
2. Allergy, sensitivity, or intolerance to the investigational product's active or inactive ingredients, or the ingredients in the standardized meals
3. Current use of hormonal contraceptives
4. Previous diagnosis of a sleep disorder or use of continuous positive air pressure (C-PAP)
5. Registered with the Canadian National Institute for the Blind (CNIB) and considered as legally blind
6. Current employment that calls for rotating shift work or shift work that will disrupt normal circadian rhythm or have worked shift work in the last 3 weeks
7. Travel across 1 or more time zones in the last 2 weeks and/or is anticipating more travel
8. Currently experiencing vivid nightmares or sleepwalking
9. Diagnosis of any pineal gland abnormalities or have undergone pinealectomy
10. Current or history of any significant diseases of the gastrointestinal tract
11. Unstable metabolic disease or chronic diseases as assessed by the QI
12. Verbal confirmation of current or pre-existing thyroid condition. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
13. Type I or Type II diabetes
14. Significant cardiovascular event in the past 6 months. Participants with no significant cardiovascular event on stable medication may be included after assessment by the QI on a case-by-case basis
15. Cancer, except skin cancers completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than 5 years after diagnosis are acceptable
16. Individuals with an autoimmune disease or are immune-compromised
17. Verbal confirmation of medical or neuropsychological condition and/or cognitive impairment that, in the QI's opinion, could interfere with study participation
18. Verbal confirmation of an HIV-, Hepatitis B- and/or C-positive diagnosis
19. History of or current diagnosis with kidney and/or liver diseases as assessed by the QI on a case-by-case basis, with the exception of history of kidney stones symptom-free for 6 months
20. Major surgery in the past 3 months or individuals who have planned surgery, that may impact the outcomes of the study, during the course of the trial. Participants will be considered on a case-by-case basis by the QI
21. Blood/bleeding disorders as determined by laboratory results
22. An acute gout attack within the past 3 months
23. Current use of prescribed medications listed in the con meds section
24. Current use of over-the-counter medications, supplements, foods and/or drinks listed in the con meds section
25. Use of medical marijuana
26. Use of recreational marijuana unless willing to undergo 1-month washout
27. Use of tobacco products within 1-year of baseline
28. Alcohol or drug abuse within the last 12 months
29. High alcohol intake (average of >2 standard drinks per day or >10 standard drinks per week)
30. Clinically significant abnormal laboratory results at screening as assessed by the QI
31. Blood donation within the past 6 months will be assessed on a case by case basis by the QI depending on volume and frequency of donation, and laboratory parameters
32. Plans to donate blood during the study or within 56 days for males and 84 days for females, the last study visit
33. Participation in other clinical research trials 30 days prior to randomization
34. Individuals who are unable to give informed consent
35. Any other active or unstable medical condition, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose a significant risk to the participant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2019-08-27 (Actual)

PRIMARY OUTCOMES:
Comparison of the pharmacokinetics of prolonged-release melatonin and immediate-release melatonin by evaluating the area under the curve (AUC 0-10h) | 7 days
Comparison of the pharmacokinetics of prolonged-release melatonin and immediate-release melatonin by evaluating the time to peak concentration (tmax) | 7 days
Comparison of the pharmacokinetics of prolonged-release melatonin and immediate-release melatonin by evaluating the peak concentration (Cmax) | 7 days
Comparison of the pharmacokinetics of prolonged-release melatonin and immediate-release melatonin by evaluating the absorption rate constant | 7 days
Comparison of the pharmacokinetics of prolonged-release melatonin and immediate-release melatonin by evaluating the elimination rate constant | 7 days
Comparison of the pharmacokinetics of prolonged-release melatonin and immediate-release melatonin by evaluating the absorption half-life | 7 days
Comparison of the pharmacokinetics of prolonged-release melatonin and immediate-release melatonin by evaluating the elimination half-life | 7 days

OTHER OUTCOMES:
Change in blood pressure after an acute administration of either prolonged-release melatonin or immediate-release melatonin | 7 days
Change in heart rate after an acute administration of either prolonged-release melatonin or immediate-release melatonin | 7 days
Change in weight after an acute administration of either prolonged-release melatonin or immediate-release melatonin | 7 days
Change in body mass index (BMI) after an acute administration of either prolonged-release melatonin or immediate-release melatonin | 7 days
Change in Red Blood Cell (RBC) count after an acute administration of either prolonged-release melatonin or immediate-release melatonin | 7 days
Change in Mean Corpuscular Volume (MCV) after an acute administration of either prolonged-release melatonin or immediate-release melatonin | 7 days
Change in Mean Corpuscular Hemoglobin (MCH) after an acute administration of either prolonged-release melatonin or immediate-release melatonin | 7 days
Change in Mean Corpuscular Hemoglobin Concentration (MCHC) after an acute administration of either prolonged-release melatonin or immediate-release melatonin | 7 days
Change in Hematocrit after an acute administration of either prolonged-release melatonin or immediate-release melatonin | 7 days
Change in Red Cell Distribution Width (RDW) after an acute administration of either prolonged-release melatonin or immediate-release melatonin | 7 days
Change in Hemoglobin (Hb) after an acute administration of either prolonged-release melatonin or immediate-release melatonin | 7 days
Change in neutrophils after an acute administration of either prolonged-release melatonin or immediate-release melatonin | 7 days
Change in lymphocytes after an acute administration of either prolonged-release melatonin or immediate-release melatonin | 7 days
Change in monocytes after an acute administration of either prolonged-release melatonin or immediate-release melatonin | 7 days
Change in eosinophils after an acute administration of either prolonged-release melatonin or immediate-release melatonin | 7 days
Change in basophils after an acute administration of either prolonged-release melatonin or immediate-release melatonin | 7 days
Change in alanine aminotransferase (ALT) after an acute administration of either prolonged-release melatonin or immediate-release melatonin | 7 days
Change in aspartate aminotransferase (AST) after an acute administration of either prolonged-release melatonin or immediate-release melatonin | 7 days
Change in creatinine after an acute administration of either prolonged-release melatonin or immediate-release melatonin | 7 days
Change in electrolytes after an acute administration of either prolonged-release melatonin or immediate-release melatonin | 7 days
  Na+, K+, and Cl- will be assessed
Change in estimated glomerular filtration rate (eGFR) after an acute administration of either prolonged-release melatonin or immediate-release melatonin | 7 days
Change in total bilirubin after an acute administration of either prolonged-release melatonin or immediate-release melatonin | 7 days
Change in adverse events after an acute administration of either prolonged-release melatonin or immediate-release melatonin | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mun JG, Wang D, Doerflein Fulk DL, Fakhary M, Gualco SJ, Grant RW, Mitmesser SH. A Randomized, Double-Blind, Crossover Study to Investigate the Pharmacokinetics of Extended-Release Melatonin Compared to Immediate-Release Melatonin in Healthy Adults. J Diet Suppl. 2024;21(2):182-194. doi: 10.1080/19390211.2023.2206475. Epub 2023 May 7. PMID 37150895